CLINICAL TRIAL: NCT00963482
Title: Secondary Prevention of Tobacco Dependence in Alcohol-dependent Patients - a Randomized, Controlled Trial
Brief Title: Smoking Cessation in Alcoholics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAG - 06.004264
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Results first posted 2012-04-13 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Smoking Cessation; Alcohol Consumption
Keywords: Smoking; Alcohol; Outcome; Harm reduction; Alcohol drinking; Treatment outcome; Treatment effectiveness
MeSH Terms: conditions — Smoking Cessation; Alcohol Drinking; Smoking; Harm Reduction | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Cognitive-behavioural smoking cessation program
  Interventions: Behavioral: Cognitive-behavioural smoking cessation program
- Control group (Other): Autogenic training
  Interventions: Behavioral: Autogenic training

INTERVENTIONS:
Behavioral: Cognitive-behavioural smoking cessation program — It's a cognitive-behavioural intervention for smoking cessation. Originally based on a 6 week program designed for outpatients (Batra & Buchkremer 2004). This program was then specifically tailored for inpatient use with additional information addressing the interaction of smoking and drinking and its consequences.
  Other Names: Nichtraucher in 6 Wochen (Batra & Buchkremer)
  Arms: Intervention group
Behavioral: Autogenic training — Learning and exercising of autogenic training. There's evidence that autogenic training is not effective in smoking cessation.
  Other Names: Autogenous Training
  Arms: Control group

SUMMARY:
Most alcohol-dependent individuals are heavy smokers. The aim of this study is to evaluate whether a specific smoking cessation program (based on cognitive-behavioral therapy) for inpatient alcohol-dependent smokers is more effective than a control condition (treatment as usual).

DETAILED DESCRIPTION:
The study is designed as a randomised, controlled trial conducted in an inpatient alcohol treatment institution. Shortly after alcohol detoxification, smokers are offered to voluntarily participate in a smoking cessation program. Participation is possible if patients either want to stop smoking or to reduce their consumption for at least 50%. Patients are asked about their smoking behaviour at the following time points: at admission (T0), after finishing the smoking cessation program or the control condition (T1), one month later by phone (T2) and six months later in a closing meeting (T3). Urine samples and CO-breath controls are taken to check both nicotine and alcohol abstinence.

ELIGIBILITY:
Inclusion Criteria:

* alcohol-dependent
* smoker
* intend to stop or reduce smoking for at least 50%

Exclusion Criteria:

* taking part in another smoking cessation program
* being pregnant
* not able to understand instruction due to cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard A. Wiesbeck, Prof. Dr., Principal Investigator — Psychiatric Hospital of the University of Basel
Locations (1):
- Psychiatric Hospital of the University of Basel, Basel, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 01.07.2007-31.01.2010 Recruiting process 31.01.2010-31.07.2011 last follow-up sessions location of recruiting: alcohol detoxification unit follow-up: outpatient
Pre-assignment Details: Out of 237 screened patients, 103 were enrolled. Intervention group(EG)=53; Control group (CG)=50.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 53 | 50
Completed | 25 | 33
Not Completed | 28 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 50 | 103
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 44 (9) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 37 | 36 | 73
Region of Enrollment [Number; unit: participants]
  Switzerland | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Smoke-free Patients
Description: Smoke-free defined with following measures:
  * patients self-report about smoking in the last 7 days (yes/no)
  * CO-level (smoke-free <10ppm)
  * urine sample (cotinine)
Time Frame: 6 months
Population: Intention-to-treat analysis
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 46 | 43
participants | 0 | 3
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; H0: "EG is equal in smoking quit rates compared to CG". H1: "EG is superior in smoking quit rates compared to CG"; Test type: Superiority or Other; p = .111, Chi-squared — not adjusted for multiple comparisons due to only two groups p<.05, two-tailed

2. Secondary Outcome: Drinking in the Last 7 Days (Patients Report + Urine Sample)
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50

LIMITATIONS AND CAVEATS:
Originally two recruiting centers were planned, what failed. Though less subjects than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No